CLINICAL TRIAL: NCT05257902
Title: Evaluation of Clinical Effectiveness of Choline Alphoscerate for Older Adults With Major Depression and Subjective Memory Complaints: a Double-blinded, Placebo-controlled, Randomization, Multicenter Investigator-initiated Trial
Brief Title: Clinical Effectiveness of Choline Alphoscerate for Older Adults With Major Depression and Subjective Memory Complaints
Acronym: CHOLDEPS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, hong jin jeon, Principal Investigator, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2021-10-033
Record Dates: First submitted 2022-01-17; First posted 2022-02-25 (Actual); Last update posted 2022-02-25 (Actual); Status verified 2022-02

CONDITIONS: Major Depression
Keywords: subjective memory complaints
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Glycerylphosphorylcholine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Active Comparator): Participants in the treatment group will take the choline alfoscerate as adjunctive therapy with their own antidepressants.
  Interventions: Drug: choline alphoscerate
- Control Group (Placebo Comparator): Participants in the control group will take the placebo, which would not affect their medical condition, for the adjunctive therapy is the choice of agreement between clinician and participants. If there is the necessity of change in antidepressant or of adjustment of their dosage, investigator can stop the clinical trial and proceed to another treatment.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: choline alphoscerate — 400mg bid/day
  Arms: Treatment group
Drug: Placebo — Placebo 1T bid/day
  Arms: Control Group

SUMMARY:
To evaluate the efficacy of choline alphoscerate on improving symptoms related to depression, anxiety, and subjective memory complaints compared to placebo in patients with Major Depressive Disorder(MDD) accompanied with subjective cognitive decline, who are over the age of 60.

DETAILED DESCRIPTION:
This clinical trial will include the participants over age 60, diagnosed as MDD under treatment of antidepressant longer than 1 month's period, assessed as Hamilton Rating Scale for Depression(HAM-D) ≥ 14, and Mini-Mental State Examination(MMSE) ≥ 20, and those who are accompanied with subjective memory complaints. The investigators will evaluate the clinical efficacy of symptomatic improvement in depression, anxiety, and subjective memory complaints. The investigators will assess these outcomes including memory function, depression, anxiety, and satisfaction on medication with scales comparing control group with treatment group under 8 weeks of medication.

This is a multi-center, randomized, double-blind, placebo-controlled, Phase IV trial to evaluate the efficacy.

Participants in the treatment group will take the choline alfoscerate as adjunctive therapy with their own antidepressants. Participants in the control group will take the placebo, which would not affect their medical condition, for the adjunctive therapy is the choice of agreement between clinician and participants. If there is the necessity of change in antidepressant or of adjustment of their dosage, investigator can stop the clinical trial and proceed to another treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 60 years
2. Diagnosed as MDD under the criteria of Diagnostic and Statistical Manual of Mental Disorders (DSM-5) and confirmed with MINI-Depression
3. HAM-D ≥ 14
4. MMSE ≥ 20
5. Who had continuous subjective memory complaints more than 6 months before the period of screening
6. Who had taking antidepressants longer than 1 month in the period of screening

Exclusion Criteria:

1. Diagnosed as schizophrenia, bipolar disorder, PTSD, OCD or other significant mental disorder under the criteria of DSM-5 (only the participants who had depressive disorder, sleep disorder, and the anxiety disorder are allowed to be included)
2. Who have medically unstable disease (only the participants, who have diabetes mellitus or hypertension under control with stable medication for 3 months could be included)
3. Diagnosed as dementia or mild cognitive impairment
4. Participants who are already taking choline alfoscerate within 6 months of period
5. Participants who have been taking medication of antipsychotics (including quetiapine), mood stabilizer, cognitive enhancer including donepezil, rivastigamine, galantamine, and memantine within 1months.
6. Participants who had previous history of liver disease or renal disease
7. Participants who had allergic reaction to choline alfoscerate
8. Other specific condition, which could be inappropriate for the trial inclusion, under the judgement of the principal investigator

Ages: 60 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-03 (Estimated); Primary Completion 2023-03 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Change of the total score of Korean version of Perceived Deficits Questionnaire-Depression | between baseline and 8weeks
  Change of the total score of Korean version of Perceived Deficits Questionnaire-Depression between the baseline and visit 5, higher scores mean a worse outcome

SECONDARY OUTCOMES:
The difference between baseline and each period of visit in the score of the first questionnaire of Memory Functioning Questionnaire (MFQ) | between baseline and each 2weeks, 4weeks, 6weeks, 8weeks
  first questionnaire of Memory Functioning Questionnaire (MFQ)
The difference between baseline and each period of visit in the score of the total Geriatric Depression Scale (GDS) | between baseline and each 2weeks, 4weeks, 6weeks, 8weeks
  total Geriatric Depression Scale (GDS), higher scores mean a worse outcome
The difference between baseline and each period of visit in the score of the Mini-Mental State Examination(MMSE) | between baseline and each 2weeks, 4weeks, 6weeks, 8weeks
  Mini-Mental State Examination(MMSE)
The difference between baseline and each period of visit in the score of the Hamilton Rating Scale for Depression(HAM-D) | between baseline and each 2weeks, 4weeks, 6weeks, 8weeks
  Hamilton Rating Scale for Depression(HAM-D), normal: 0~6 score, mild: 7~18 score, moderate: 18-24 score, severe: above 25 score
The difference between baseline and each period of visit in the score of the Hamilton Rating Scale for Anxiety (HAM-A) | between baseline and each 2weeks, 4weeks, 6weeks, 8weeks
  Hamilton Rating Scale for Anxiety (HAM-A), mild: below17 score, moderate: 18-24 score, severe: above 30 score
The difference the score | between baseline and each 2weeks, 4weeks, 6weeks, 8weeks
  The difference between baseline and each period of visit in the score of the Korea version of montreal cognitive assessment (K-MoCA)
The difference between baseline and each period of visit in the score of the total score of Medication Satisfaction Questionnaire (MSQ) | between baseline and each 2weeks, 4weeks, 6weeks, 8weeks
  total score of Medication Satisfaction Questionnaire (MSQ)
assessement AE | between baseline and each 2weeks, 4weeks, 6weeks, 8weeks
  collected all Adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Hong Jin JEON, Principal Investigator — Samsung Medical Center